CLINICAL TRIAL: NCT02516241
Title: A Phase III, Randomized, Open-Label, Controlled, Multi-Center, Global Study of First-Line MEDI4736 (Durvalumab) Monotherapy and MEDI4736 (Durvalumab) in Combination With Tremelimumab Versus Standard of Care Chemotherapy in Patients With Unresectable Stage IV Urothelial Cancer
Brief Title: Study of MEDI4736 (Durvalumab) With or Without Tremelimumab Versus Standard of Care Chemotherapy in Urothelial Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419BC00001; 2015-001633-24 (EudraCT Number)
Record Dates: First submitted 2015-07-13; First posted 2015-08-05 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Cancer
Keywords: Urothelial Cancer; Phase III
MeSH Terms: interventions — durvalumab; tremelimumab; Cisplatin; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combination Therapy (Experimental): MEDI4736 (Durvalumab) + Tremelimumab
  Interventions: Drug: MEDI4736 (Durvalumab); Drug: Tremelimumab
- Monotherapy (Experimental): MEDI4736 (Durvalumab)
  Interventions: Drug: MEDI4736 (Durvalumab)
- Standard of Care (Active Comparator): Standard of Care Chemotherapy Treatment
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: MEDI4736 (Durvalumab) — IV infusion
  Arms: Combination Therapy; Monotherapy
Drug: Tremelimumab — IV infusion
  Arms: Combination Therapy
Drug: Cisplatin — IV infusion
  Arms: Standard of Care
Drug: Carboplatin — IV infusion
  Arms: Standard of Care
Drug: Gemcitabine — IV infusion
  Arms: Standard of Care

SUMMARY:
A Phase III, Randomized, Open-Label, Controlled, Multi-Center, Global Study of First-Line MEDI4736 (Durvalumab) Monotherapy and MEDI4736 (Durvalumab) in Combination with Tremelimumab Versus Standard of Care Chemotherapy in Patients with Stage IV Urothelial Cancer

DETAILED DESCRIPTION:
This is a randomized, open-label, controlled, multi-center, global Phase III study to determine the efficacy and safety of MEDI4736 (Durvalumab) monotherapy and MEDI4736 (Durvalumab) in combination with tremelimumab versus SoC (cisplatin + gemcitabine or carboplatin + gemcitabine doublet) first-line chemotherapy in treatment-naïve patients with histologically or cytologically documented, unresectable, Stage IV transitional cell carcinoma (transitional cell and mixed transitional/non-transitional cell histologies) of the urothelium (including renal pelvis, ureters, urinary bladder, and urethra) and to allow sufficient flexibility for Investigators and patients to select the agents that reflect their normal clinical practice and national guidelines. The patients enrolled in the study will be randomized 1:1:1 to receive treatment with combination therapy, monotherapy, or SoC (cisplatin + gemcitabine or carboplatin + gemcitabine, based on cisplatin eligibility). Patients will be treated with MEDI4736 (Durvalumab) or MEDI4736 (Durvalumab) with tremelimumab, or treated with SoC until progressive disease (PD) is confirmed, unacceptable toxicity occurs, withdrawal of consent, or another discontinuation criterion is met. Patients will be followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically documented, unresectable, Stage IV transitional cell carcinoma of the urothelium who have not been previously treated with first-line chemotherapy.
* Patients eligible or ineligible for cisplatin-based chemotherapy. Cisplatin ineligibility is defined as meeting 1 of the following criteria: • Creatinine clearance (calculated or measured) <60 mL/min calculated by Cockcroft-Gault equation (using actual body weight) or by measured 24-hour urine collection for determination • Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 audiometric hearing loss • CTCAE Grade ≥2 peripheral neuropathy • New York Heart Association ≥Class III heart failure.
* Tumor PD-L1 status, with Immunohistochemical (IHC) assay confirmed by a reference laboratory, must be known prior to randomization.

Exclusion Criteria:

* Prior exposure to immune-mediated therapy, including but not limited to, other anti cytotoxic T-lymphocyte-associated protein 4 (CTLA 4), anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies, including therapeutic anticancer vaccines. Prior local intervesical chemotherapy or immunotherapy is allowed if completed at least 28 days prior to the initiation of study treatment.
* History of allogenic organ transplantation that requires use of immunosuppressive agents.
* Active or prior documented autoimmune or inflammatory disorders. The following are exceptions to this criterion: • Patients with vitiligo or alopecia • Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement • Any chronic skin condition that does not require systemic therapy • Patients without active disease in the last 3 years may be included but only after consultation with AstraZeneca • Patients with celiac disease controlled by diet alone may be included but only after consultation with AstraZeneca.
* Brain metastases or spinal cord compression unless the patient's condition is stable and off steroids for at least 14 days prior to the start of study treatment. Patients with suspected or known brain metastases at screening should have an MRI (preferred)/CT, preferably with IV contrast to access baseline disease status.
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of investigational product (IP). The following are exceptions to this criterion: • Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection) • Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent • Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IP.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1126 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (181):
- United States (15):
  - Research Site, Los Angeles, California
  - Research Site, Stanford, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, New York, New York
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Seattle, Washington
- Australia (5):
  - Research Site, Box Hill
  - Research Site, Elizabeth Vale
  - Research Site, Macquarie University
  - Research Site, St Leonards
  - Research Site, Waratah
- Austria (2):
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Ijuí
  - Research Site, Itajaí
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- China (11):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Xi'an
  - Research Site, Xiamen
- Denmark (4):
  - Research Site, Århus C
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Odense C
- France (9):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Suresnes
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (7):
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, München
  - Research Site, Münster
- Greece (6):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Holargos, Athens
  - Research Site, Maroussi, Athens
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Ẕerifin
- Italy (8):
  - Research Site, Arezzo
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo
- Japan (28):
  - Research Site, Akita
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hakata-shi
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Izumo-shi
  - Research Site, Kagoshima
  - Research Site, Kanazawa
  - Research Site, Kita-gun
  - Research Site, Kobe
  - Research Site, Koshigaya-shi
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Morioka
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Saga
  - Research Site, Sagamihara-shi
  - Research Site, Sakura-shi
  - Research Site, Sapporo
  - Research Site, Suita-shi
  - Research Site, Takatsuki-shi
  - Research Site, Yokohama
- Mexico (5):
  - Research Site, Guadalajara
  - Research Site, León
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
- Netherlands (7):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Enschede
  - Research Site, Groningen
  - Research Site, Leiden
  - Research Site, Maastricht
  - Research Site, Nijmegen
- Poland (7):
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Gliwice
  - Research Site, Olsztyn
  - Research Site, Otwock
  - Research Site, Szczecin
  - Research Site, Warsaw
- Portugal (3):
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Porto
- Russia (8):
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Nizhnyi Novgorod
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Yaroslavl
- South Korea (3):
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, Badajoz
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Elche(Alicante)
  - Research Site, Madrid
  - Research Site, Pozuelo de Alarcón
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Izmir
- United Kingdom (9):
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Sheffield
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Powles T, van der Heijden MS, Castellano D, Galsky MD, Loriot Y, Petrylak DP, Ogawa O, Park SH, Lee JL, De Giorgi U, Bogemann M, Bamias A, Eigl BJ, Gurney H, Mukherjee SD, Fradet Y, Skoneczna I, Tsiatas M, Novikov A, Suarez C, Fay AP, Duran I, Necchi A, Wildsmith S, He P, Angra N, Gupta AK, Levin W, Bellmunt J; DANUBE study investigators. Durvalumab alone and durvalumab plus tremelimumab versus chemotherapy in previously untreated patients with unresectable, locally advanced or metastatic urothelial carcinoma (DANUBE): a randomised, open-label, multicentre, phase 3 trial. Lancet Oncol. 2020 Dec;21(12):1574-1588. doi: 10.1016/S1470-2045(20)30541-6. Epub 2020 Sep 21. PMID 32971005
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419BC00001&attachmentIdentifier=bfebc14d-a0f4-45b7-89cb-4a165e27074b&fileName=D419BC00001_SAPv5-redacted.pdf&versionIdentifier=
- See also: Redacted Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419BC00001&attachmentIdentifier=a04d44be-8078-4bc2-9423-9816fa57e99d&fileName=d419bc00001-CSP-v9-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Started | 342 | 346 | 344
Received Treatment | 340 | 345 | 313
Completed | 0 | 0 | 0
Not Completed | 342 | 346 | 344
Not completed — Death | 255 | 262 | 270
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 7 | 12
Not completed — participants ongoing at data cut-off | 84 | 76 | 59

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy | Monotherapy | Standard of Care | Total
Number analyzed (Participants) | 342 | 346 | 344 | 1032
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 66.4 (9.60) | 66.3 (9.9) | 67.0 (9.32) | 66.5 (9.60)
Age, Customized [Count of Participants; unit: Participants]
  Age Group (Years): <50 | 19 | 22 | 14 | 55
  Age Group (Years): >= 50 - < 65 | 118 | 115 | 119 | 352
  Age Group (Years): >= 65 - < 75 | 132 | 141 | 137 | 410
  Age Group (Years): >= 75 | 73 | 68 | 74 | 215
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 86 | 97 | 70 | 253
  Sex: Male | 256 | 249 | 274 | 779
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 15 | 14 | 17 | 46
  Ethnicity: Not Hispanic or Latino | 320 | 329 | 322 | 971
  Ethnicity: Unknown or Not Reported | 7 | 3 | 5 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 253 | 278 | 260 | 791
  Race: Black or African American | 3 | 3 | 0 | 6
  Race: Asian | 72 | 60 | 76 | 208
  Race: Native Hawaiian or other Pacific islander | 0 | 0 | 0 | 0
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Other | 13 | 4 | 8 | 25
  Race: Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Efficacy of Durvalumab + Tremelimumab Combination Therapy Versus SoC in Terms of OS in Full Analysis Set
Description: The OS was defined as the time from the date of randomization until death due to any cause (ie, date of death or censoring - date of randomization + 1). Any participant not known to have died at the time of analysis were censored based on the last recorded date on which the participant was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
Time Frame: From randomization date until death due to any cause, assessed up to the data cut-off date (27JAN2020, a maximum of 5 years).
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Standard of Care
Number analyzed (Participants) | 342 | 344
Months | 15.1 [13.1 to 18.0] | 12.1 [10.9 to 14]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.0751, Log Rank — The 2-sided p-value was calculated using a stratified log-rank test adjusting for PD-L1 status, visceral metastases and cisplatin eligibility status; Hazard Ratio (HR) = 0.85, 98.66% CI 2-sided [0.688 to 1.063] — The HR and confidence interval (CI) were calculated using a stratified Cox proportional hazards model, adjusting for PD-L1 status, visceral metastases and cisplatin eligibility status with ties handled by the Breslow approach

2. Primary Outcome: To Assess the Efficacy of Durvalumab Monotherapy Versus SoC in Terms of OS in PD-L1-High Analysis Set
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PD-L1-High analysis set will include the subset of patients in the FAS whose PD-L1 status is PD-L1-High as defined by an Immunohistochemistry (IHC) assay developed by Ventana as:
  ≥25% tumor cell membrane positivity for PD-L1 at any intensity above background staining as noted on the corresponding negative control OR ≥25% tumor associated immune cell positivity for PD-L1 at any intensity above background staining as noted on the corresponding negative control
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Monotherapy | Standard of Care
Number analyzed (Participants) | 209 | 207
Months | 14.4 [10.4 to 17.3] | 12.1 [10.4 to 15.0]
Statistical Analysis 1: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p = 0.3039, Log Rank — The 2-sided p-value was calculated using a stratified log-rank test adjusting for visceral metastases and cisplatin eligibility status; Hazard Ratio (HR) = 0.89, 96.99% CI 2-sided [0.695 to 1.139] — The HR and confidence interval (CI) were calculated using a stratified Cox proportional hazards model, adjusting for visceral metastases and cisplatin eligibility status with ties handled by the Breslow approach

3. Secondary Outcome: OS, Full Analysis Set - Durvalumab Monotherapy vs SoC
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Monotherapy | Standard of Care
Number analyzed (Participants) | 346 | 344
Months | 13.2 [10.3 to 15] | 12.1 [10.9 to 14]
Statistical Analysis 1: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p = 0.8637, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.830 to 1.169] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: OS, PD-L1-High Analysis Set -Durvalumab + Tremelimumab Combination Therapy Versus SoC
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Standard of Care
Number analyzed (Participants) | 205 | 207
Months | 17.9 [14.8 to 24.2] | 12.1 [10.4 to 15.0]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.0091, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.589 to 0.928] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: OS, PD-L1-Low/Negative Analysis Set -Durvalumab + Tremelimumab Combination Therapy Versus SoC and Durvalumab + Tremelimumab Combination Therapy Versus Durvalumab Monotherapy
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PD-L1-Low/Negative analysis set will include the subset of patients in the FAS whose PD-L1 status is PD-L1-Low/negative as defined by an Immunohistochemistry (IHC) assay developed by Ventana as:
  <25% tumor cell membrane positivity for PD-L1 at any intensity above background staining as noted on the corresponding negative control AND <25% tumor associated immune cell positivity for PD-L1 at any intensity above background staining as noted on the corresponding negative control.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
Months | 11.8 [8.9 to 15.8] | 10.9 [8.0 to 14.8] | 12.2 [10.4 to 14]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.7599, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.799 to 1.359] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Combination Therapy vs Monotherapy; monotherapy as reference; Test type: Superiority; p = 0.4424, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.692 to 1.175] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Alive at 24 Months (OS24), Full Analysis Set
Description: Alive at 24 months (OS24) is defined as the Kaplan-Meier estimate of OS at 24 months.
Time Frame: From randomization date until death due to any cause, assessed up to 24 months or the data cut-off date (27JAN2020).
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
percentage of participants | 39.0 [33.8 to 44.2] | 31.5 [26.6 to 36.4] | 29.0 [24.2 to 34.0]

7. Secondary Outcome: Alive at 24 Months (OS24), PD-L1-High Analysis Set
Description: Alive at 24 months (OS24) is defined as the Kaplan-Meier estimate of OS at 24 months.
Time Frame: From randomization date until death due to any cause, assessed up to 24 months or the data cut-off date (27JAN2020).
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
percentage of participants | 43.7 [36.8 to 50.3] | 36.0 [29.5 to 42.6] | 29.3 [23.1 to 35.7]

8. Secondary Outcome: Alive at 24 Months (OS24), PD-L1-Low/Negative Analysis Set
Description: Alive at 24 months (OS24) is defined as the Kaplan-Meier estimate of OS at 24 months.
Time Frame: From randomization date until death due to any cause, assessed up to 24 months or the data cut-off date (27JAN2020).
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
percentage of participants | 32.1 [24.5 to 40.0] | 24.5 [17.6 to 32.0] | 28.6 [21.2 to 36.4]

9. Secondary Outcome: PFS, Full Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: Progression free survival (PFS) (per RECIST 1.1, as assessed by investigator) was defined as the time from the date of randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from randomized therapy or receives another anticancer therapy prior to progression.
  Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at baseline then every 8 weeks since randomization until confirmed disease progression. Assessed up to the data cut-off date (27JAN2020, a maximum of 5 years).
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
Months | 3.7 [3.4 to 3.8] | 2.3 [1.9 to 3.5] | 6.7 [5.7 to 7.3]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.2579, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.931 to 1.304] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p = 0.0008, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [1.124 to 1.567] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: PFS, PD-L1-High Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Monotherapy vs SoC
Description: as for outcome 9
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
Months | 4.1 [3.6 to 5.7] | 2.4 [1.9 to 3.7] | 5.8 [5.6 to 7.2]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.2395, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.705 to 1.091] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p = 0.2431, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.917 to 1.406] — [estimate comment as in outcome 2, analysis 1]

11. Secondary Outcome: PFS, PD-L1-Low/Negative Analysis Set -Durvalumab + Tremelimumab Combination Therapy Versus SoC and Durvalumab + Tremelimumab Combination Therapy Versus Durvalumab Monotherapy
Description: as for outcome 9
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
Months | 2.0 [1.9 to 3.6] | 2.0 [1.9 to 3.5] | 7.2 [5.7 to 7.5]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.0014, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.53, 95% CI 2-sided [1.177 to 1.990] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Combination Therapy vs Monotherapy; monotherapy as reference; Test type: Superiority; p = 0.6236, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.729 to 1.209] — [estimate comment as in outcome 2, analysis 1]

12. Secondary Outcome: Alive and Progression-free at 12 Months (APF12), Full Analysis Set
Description: Alive and progression-free at 12 months (APF12) was defined as the Kaplan-Meier estimate of PFS (per RECIST 1.1 as assessed by investigator) at 12 months.
Time Frame: Tumour scans performed at baseline then every 8 weeks since randomization until confirmed disease progression. Assessed up to 12 months or the data cut-off date (27JAN2020).
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
percentage of participants | 21.4 [17.2 to 26.0] | 16.8 [13.1 to 21.1] | 15.3 [11.4 to 19.7]

13. Secondary Outcome: Alive and Progression-free at 12 Months (APF12), PD-L1-High Analysis Set
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
percentage of participants | 25.6 [19.7 to 31.8] | 21.2 [15.9 to 27.0] | 15.0 [10.2 to 20.7]

14. Secondary Outcome: Alive and Progression-free at 12 Months (APF12), PD-L1-Low/Negative Analysis Set
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
percentage of participants | 15.2 [9.6 to 21.8] | 9.7 [5.4 to 15.7] | 15.6 [9.6 to 22.9]

15. Secondary Outcome: PFS2, Full Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: Time from randomization to second progression or death (PFS2) was defined as the time from the date of randomization to the earliest of the progression event subsequent to first subsequent therapy or death (ie, date of PFS2 event or censoring - date of randomization +1).
  Median PFS2 was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at baseline then every 8 weeks since randomization until first confirmed disease progression, disease then assessed per local practice until 2nd progression. Assessed up to the data cut-off date (27JAN2020, a maximum of 5 years).
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
Months | 14.6 [11.3 to 17.8] | 11.9 [8.9 to 14.6] | 11.5 [10.3 to 12.8]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.0477, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.683 to 0.998] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p = 0.7885, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.809 to 1.175] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: PFS2, PD-L1-High Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Monotherapy vs SoC
Description: as for outcome 15
Time Frame: as for outcome 15
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
Months | 17.2 [12.1 to 24.8] | 13.4 [9.7 to 17.5] | 11.3 [8.9 to 14.3]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.0053, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.549 to 0.901] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p = 0.1336, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.651 to 1.059] — [estimate comment as in outcome 2, analysis 1]

17. Secondary Outcome: PFS2, PD-L1-Low/Negative Analysis Set -Durvalumab + Tremelimumab Combination Therapy Versus SoC and Durvalumab + Tremelimumab Combination Therapy Versus Durvalumab Monotherapy
Description: as for outcome 15
Time Frame: as for outcome 15
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
Months | 10.7 [7.5 to 16.6] | 9.4 [7.0 to 13.7] | 11.6 [10.3 to 13.4]
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.8148, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.772 to 1.391] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Combination Therapy vs Monotherapy; monotherapy as reference; Test type: Superiority; p = 0.2684, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.636 to 1.134] — [estimate comment as in outcome 2, analysis 1]

18. Secondary Outcome: Objective Response Rate (ORR), Full Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: Objective response rate ORR (per RECIST 1.1 as assessed by investigator) is defined as the number (%) of patients with at least 1 visit response of CR or PR.
Time Frame: as for outcome 9
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
percentage of participants | 36.3 | 25.7 | 49.1
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.0005, Regression, Logistic — P-value was based on twice the change in log-likelihood resulting from logistic regression model, adjusting for PD-L1 status, visceral metastases and cisplatin eligibility status; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.422 to 0.788] — The OR and confidence interval (CI) were calculated using logistic regression, adjusting for PD-L1 status, visceral metastases and cisplatin eligibility status
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.253 to 0.485] — [estimate comment as in outcome 18, analysis 1]

19. Secondary Outcome: Objective Response Rate (ORR), PD-L1-High Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Monotherapy vs SoC
Description: as for outcome 18
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
percentage of participants | 46.8 | 27.8 | 48.3
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.7708, Regression, Logistic — P-value was based on twice the change in log-likelihood resulting from logistic regression model, adjusting for visceral metastases and cisplatin eligibility status; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.639 to 1.394] — The OR and confidence interval (CI) were calculated using logistic regression, adjusting for visceral metastases and cisplatin eligibility status
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.268 to 0.610] — [estimate comment as in outcome 19, analysis 1]

20. Secondary Outcome: Objective Response Rate (ORR), PD-L1-Low/Negative Analysis Set -Durvalumab + Tremelimumab Combination Therapy Versus SoC and Durvalumab + Tremelimumab Combination Therapy Versus Durvalumab Monotherapy
Description: as for outcome 18
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
percentage of participants | 20.4 | 22.6 | 50.4
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.135 to 0.406] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: Combination Therapy vs Monotherapy; monotherapy as reference; Test type: Superiority; p = 0.6195, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.469 to 1.566] — [estimate comment as in outcome 19, analysis 1]

21. Secondary Outcome: Objective Response Rate (ORR) Based on BICR Assessment According to RECIST 1.1 - Responses Are Confirmed - Durvalumab Cisplatin Ineligible Population
Description: Objective response rate ORR (per RECIST 1.1 as assessed by investigator) is defined as the number (%) of patients with at least 1 visit response of CR or PR.
  unconfirmed responses are excluded.
Time Frame: Tumour scans performed at baseline then every 8 weeks since randomization until confirmed disease progression. Assessed up to the data cut-off date (01NOV2017, a maximum of 3 years).
Population: Durvalumab Cisplatin Ineligible Population include all patients who had received D monotherapy and were not eligible for cisplatin treatment at baseline (per eCRF).
Measure: Number; unit: percentage of participants
Groups:
- Monotherapy - PD-L1 High: MEDI4736 (Durvalumab) - PD-L1 high
- Monotherapy - PD-L1 Low/Negative: MEDI4736 (Durvalumab) - PD-L1 low/negative
- Monotherapy - Total: MEDI4736 (Durvalumab)
Arm/Group | Monotherapy - PD-L1 High | Monotherapy - PD-L1 Low/Negative | Monotherapy - Total
Number analyzed (Participants) | 87 | 56 | 143
percentage of participants | 23.0 | 17.9 | 21.0

22. Secondary Outcome: Disease Control Rate (DCR) at 6 Months, Full Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: Disease control rate (DCR) at 6 months is defined as the percentage of patients who have a best objective response (BoR) of CR or PR, or who have demonstrated SD for a minimum interval of 24 weeks (-7 days, i.e., 161 days), following the start of study treatment.
Time Frame: Tumour scans performed at baseline then every 8 weeks since randomization until confirmed disease progression. Assessed up to 6 months or the data cut-off date (27JAN2020).
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
percentage of participants | 41.5 | 31.8 | 55.5
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.410 to 0.759] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.267 to 0.500] — [estimate comment as in outcome 18, analysis 1]

23. Secondary Outcome: Disease Control Rate (DCR) at 6 Months, PD-L1-High Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Monotherapy vs SoC
Description: as for outcome 22
Time Frame: as for outcome 22
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
percentage of participants | 49.8 | 34.4 | 53.1
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.4959, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.590 to 1.291] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.305 to 0.679] — [estimate comment as in outcome 19, analysis 1]

24. Secondary Outcome: Disease Control Rate (DCR) at 6 Months, PD-L1-Low/Negative Analysis Set -Durvalumab + Tremelimumab Combination Therapy Versus SoC and Durvalumab + Tremelimumab Combination Therapy Versus Durvalumab Monotherapy
Description: as for outcome 22
Time Frame: as for outcome 22
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
percentage of participants | 29.2 | 27.7 | 59.1
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.160 to 0.448] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: Combination Therapy vs Monotherapy; monotherapy as reference; Test type: Superiority; p = 0.8074, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.623 to 1.836] — [estimate comment as in outcome 19, analysis 1]

25. Secondary Outcome: Disease Control Rate (DCR) at 12 Months, Full Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: Disease control rate (DCR) at 12 months is defined as the percentage of patients who have a best objective response (BoR) of CR or PR, or who have demonstrated SD for a minimum interval of 48 weeks (-7 days, i.e., 329 days), following the start of study treatment.
Time Frame: as for outcome 12
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
percentage of participants | 38.0 | 28.0 | 50.6
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.0008, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.432 to 0.802] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.270 to 0.512] — [estimate comment as in outcome 18, analysis 1]

26. Secondary Outcome: Disease Control Rate (DCR) at 12 Months, PD-L1-High Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Monotherapy vs SoC
Description: as for outcome 25
Time Frame: as for outcome 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
percentage of participants | 47.3 | 30.6 | 48.8
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p = 0.7717, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.639 to 1.394] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.303 to 0.682] — [estimate comment as in outcome 19, analysis 1]

27. Secondary Outcome: Disease Control Rate (DCR) at 12 Months, PD-L1-Low/Negative Analysis Set -Durvalumab + Tremelimumab Combination Therapy Versus SoC and Durvalumab + Tremelimumab Combination Therapy Versus Durvalumab Monotherapy
Description: as for outcome 25
Time Frame: as for outcome 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
percentage of participants | 24.1 | 24.1 | 53.3
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.151 to 0.439] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: Combination Therapy vs Monotherapy; monotherapy as reference; Test type: Superiority; p = 0.9692, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.556 to 1.759] — [estimate comment as in outcome 19, analysis 1]

28. Secondary Outcome: Duration of Response (DoR), Full Analysis Set
Description: Duration of response (DoR) (per RECIST 1.1 as assessed by investigator) was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression (i.e. date of PFS event or censoring - date of first response + 1).
Time Frame: as for outcome 9
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
Months | 11.1 [4.3 to NA] — upper limit is not reached | 9.3 [5.4 to NA] — upper limit is not reached | 5.7 [3.7 to 9.3]

29. Secondary Outcome: Duration of Response (DoR), PD-L1-High Analysis Set
Description: as for outcome 28
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
Months | 10.0 [3.8 to NA] — upper limit is not reached. | 18.5 [5.6 to NA] — upper limit is not reached. | 5.8 [3.7 to 11.5]

30. Secondary Outcome: Duration of Response (DoR), PD-L1-Low/Negative Analysis Set
Description: as for outcome 28
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
Months | 12.9 [5.5 to NA] — upper limit is not reached. | 5.6 [3.8 to NA] — upper limit is not reached. | 5.7 [3.9 to 8.2]

31. Secondary Outcome: Serum Concentrations of Durvalumab, Pharmacokinetic Analysis Set
Description: Blood samples were collected to determine the serum concentration of durvalumab.
Time Frame: Pre-dose and within 1 hour after end of infusion at Week 0, 12 and 24, pre-dose at week 4, and at follow-up Month 3.
Population: Pharmacokinetic analysis set included all patients who received at least 1 dose of durvalumab or tremelimumab per the protocol and had at least one post dose evaluable PK data of durvalumab or tremelimumab
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Combination Therapy | Monotherapy
Number analyzed (Participants) | 339 | 343
μg/mL
  Week 0 - Predose: number analyzed (Participants) | 329 | 339
  Week 0 - Predose | NA (NA) — week 0 pre-dose serum concentrations are below the level of detection | NA (NA) — week 0 pre-dose serum concentrations are below the level of detection
  Week 0 - Postdose: number analyzed (Participants) | 328 | 334
  Week 0 - Postdose | 511 (338) | 484 (162)
  Week 4 - Predose: number analyzed (Participants) | 285 | 300
  Week 4 - Predose | 75.3 (84.4) | 78.9 (56.5)
  Week 12 - Predose: number analyzed (Participants) | 198 | 195
  Week 12 - Predose | 125 (97.7) | 144 (82.5)
  Week 12 - Postdose: number analyzed (Participants) | 184 | 186
  Week 12 - Postdose | 594 (298) | 576 (233)
  Week 24 - Predose: number analyzed (Participants) | 127 | 119
  Week 24 - Predose | 150 (94.4) | 163 (82.5)
  Week 24 - Postdose: number analyzed (Participants) | 126 | 116
  Week 24 - Postdose | 604 (249) | 600 (244)
  Follow-up Month 3: number analyzed (Participants) | 77 | 66
  Follow-up Month 3 | 23.3 (50) | 19.9 (18.4)

32. Secondary Outcome: Serum Concentrations of Tremelimumab, Pharmacokinetic Analysis Set
Description: Blood samples were collected to determine the serum concentration of tremelimumab.
Time Frame: Pre-dose and within 1 hour after end of infusion at Week 0, 12 and 24, pre-dose at week 4, and at follow-up Month 3.
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Combination Therapy
Number analyzed (Participants) | 339
μg/mL
  Week 0 - Predose: number analyzed (Participants) | 332
  Week 0 - Predose | NA (NA) — week 0 pre-dose serum concentrations are below the level of detection
  Week 0 - Postdose: number analyzed (Participants) | 332
  Week 0 - Postdose | 24.0 (11.5)
  Week 4 - Predose: number analyzed (Participants) | 283
  Week 4 - Predose | 3.75 (3.18)
  Week 12 - Predose: number analyzed (Participants) | 197
  Week 12 - Predose | 5.43 (4.01)
  Week 12 - Postdose: number analyzed (Participants) | 182
  Week 12 - Postdose | 28.1 (13.2)
  Follow-up Month 3: number analyzed (Participants) | 63
  Follow-up Month 3 | 0.943 (1.40)

33. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Durvalumab, Safety Analysis Set - ADA Evaluable Patients
Description: Serum Samples will be measured for the presence of ADAs and ADA-neutralizing antibodies for Durvalumab using validated assays. Tiered analysis will be performed to include screening, confirmatory, and titer assay components, and positive-negative cut points previously statistically determined from drug-naïve validation samples will be used. Persistently positive is defined as having at least 2 post-baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. Transiently positive is defined as having at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. The category may include patients meeting these criteria who are ADA positive at baseline.
Time Frame: At week 0, 4, 12 and 24, and at follow-up Month 3.
Population: ADA evaluable patients is defined as patients in the safety analysis set who have a non-missing baseline ADA and at least one non-missing post-baseline result
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy | Monotherapy
Number analyzed (Participants) | 340 | 345
Participants
  ADA evaluable patients | 293 | 302
  ADA positive at any visit (ADA Prevalence): number analyzed (Participants) | 293 | 302
  ADA positive at any visit (ADA Prevalence) | 37 | 31
  Treatment-emergent ADA positive (ADA Incidence): number analyzed (Participants) | 293 | 302
  Treatment-emergent ADA positive (ADA Incidence) | 28 | 11
  Treatment-boosted ADA: number analyzed (Participants) | 293 | 302
  Treatment-boosted ADA | 0 | 1
  Treatment-induced ADA (Positive Post-baseline only): number analyzed (Participants) | 293 | 302
  Treatment-induced ADA (Positive Post-baseline only) | 28 | 10
  ADA Positive at Baseline only: number analyzed (Participants) | 293 | 302
  ADA Positive at Baseline only | 8 | 18
  ADA Positive Post-baseline and Positive at Baseline: number analyzed (Participants) | 293 | 302
  ADA Positive Post-baseline and Positive at Baseline | 1 | 3
  Persistently Positive: number analyzed (Participants) | 293 | 302
  Persistently Positive | 15 | 8
  Transiently Positive: number analyzed (Participants) | 293 | 302
  Transiently Positive | 14 | 5
  nAb Positive at any visit: number analyzed (Participants) | 293 | 302
  nAb Positive at any visit | 3 | 2

34. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Tremelimumab, Safety Analysis Set - ADA Evaluable Patients
Description: Serum Samples will be measured for the presence of ADAs and ADA-neutralizing antibodies for Tremelimumab using validated assays. Tiered analysis will be performed to include screening, confirmatory, and titer assay components, and positive-negative cut points previously statistically determined from drug-naïve validation samples will be used. Persistently positive is defined as having at least 2 post-baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. Transiently positive is defined as having at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. The category may include patients meeting these criteria who are ADA positive at baseline.
Time Frame: At week 0, 4, 12 and at follow-up Month 3.
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 340
Participants
  ADA evaluable patients | 292
  ADA positive at any visit (ADA Prevalence): number analyzed (Participants) | 292
  ADA positive at any visit (ADA Prevalence) | 64
  Treatment-emergent ADA positive (ADA Incidence): number analyzed (Participants) | 292
  Treatment-emergent ADA positive (ADA Incidence) | 54
  Treatment-boosted ADA: number analyzed (Participants) | 292
  Treatment-boosted ADA | 1
  Treatment-induced ADA (Positive Post-baseline only): number analyzed (Participants) | 292
  Treatment-induced ADA (Positive Post-baseline only) | 53
  ADA Positive at Baseline only: number analyzed (Participants) | 292
  ADA Positive at Baseline only | 8
  ADA Positive Post-baseline and Positive at Baseline: number analyzed (Participants) | 292
  ADA Positive Post-baseline and Positive at Baseline | 3
  Persistently Positive: number analyzed (Participants) | 292
  Persistently Positive | 31
  Transiently Positive: number analyzed (Participants) | 292
  Transiently Positive | 25
  nAb Positive at any visit: number analyzed (Participants) | 292
  nAb Positive at any visit | 50

35. Secondary Outcome: Change From Baseline in FACT-BL (Derived NFBlSI-18 Score, FACT-BL TOI, and FACT-BL Total Score) by MMRM Analysis, Full Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: the change from baseline in the following total/index scores will be evaluated as secondary endpoints: FACT-BL TOI (refer to as TOI), FACT-BL Total score, and NFBlSI-18 score.
  All the 5 subscales (PWB (0-28), FWB (0-28), EWB (0-24), SWB (0-28), and BlCS(0-48)) are summed as the FACT-BL total score (range 0-156), while the sum of PWB, FWB and BICS constitutes the FACT-BL TOI (range 0-104).
  NFBlSI-18 (range 0-72) is based on the scores of 16 items (GP4, C2, BL1, GP3, GE6, GE1, C6, BL5, GF5, GP2, GP1, GP6, C3, GP5, GF3, GF7) and 2 extra items "I feel weak all overall" and "I feel light-headed (dizzy)". The range of each item is 0-4.
  Higher score represent worse outcome.
Time Frame: At baseline then every 8 weeks until second progression/death, whichever comes first. Assessed up to the data cut-off date (27JAN2020, a maximum of 5 years).
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
Scores on a scale
  NFBLSI - 18 Score (Average overall visits): number analyzed (Participants) | 220 | 204 | 189
  NFBLSI - 18 Score (Average overall visits) | -3.7 (0.70) | -3.1 (0.76) | -5.2 (0.82)
  FACT-BL TOI (Average overall visits): number analyzed (Participants) | 220 | 204 | 189
  FACT-BL TOI (Average overall visits) | -5.5 (0.87) | -3.9 (0.95) | -7.2 (1.02)
  FACT-BL Total score (Average overall visits): number analyzed (Participants) | 220 | 204 | 189
  FACT-BL Total score (Average overall visits) | -7.2 (1.19) | -4.7 (1.30) | -8.8 (1.39)
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; NFBLSI- 18 score (Average overall visits); Test type: Superiority; p = 0.1617, Mixed Models Analysis — MMRM model included patient, treatment, cisplatin eligibility, PD-L1 status and visceral metastasis, visit and treatment by visit interaction as explanatory variables, and the appropriate baseline FACT-BL value as a covariate; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.6 to 3.59]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; NFBLSI- 18 score (Average overall visits); Test type: Superiority; p = 0.0578, Mixed Models Analysis — [p-value comment as in outcome 35, analysis 1]; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-0.07 to 4.29]
Statistical Analysis 3: Comparison: Combination Therapy vs Standard of Care; FACT-BL TOI (Average overall visits); Test type: Superiority; p = 0.2003, Mixed Models Analysis — [p-value comment as in outcome 35, analysis 1]; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-0.91 to 4.32]
Statistical Analysis 4: Comparison: Monotherapy vs Standard of Care; FACT-BL TOI (Average overall visits); Test type: Superiority; p = 0.0178, Mixed Models Analysis — [p-value comment as in outcome 35, analysis 1]; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [0.57 to 6.00]
Statistical Analysis 5: Comparison: Combination Therapy vs Standard of Care; FACT-BL Total score (Average overall visits); Test type: Superiority; p = 0.3765, Mixed Models Analysis — [p-value comment as in outcome 35, analysis 1]; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-1.96 to 5.17]
Statistical Analysis 6: Comparison: Monotherapy vs Standard of Care; FACT-BL Total score (Average overall visits); Test type: Superiority; p = 0.0300, Mixed Models Analysis — [p-value comment as in outcome 35, analysis 1]; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [0.40 to 7.81]

36. Secondary Outcome: Change From Baseline in FACT-BL (Derived NFBlSI-18 Score, FACT-BL TOI, and FACT-BL Total Score) by MMRM Analysis, PD-L1-High Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: the change from baseline in the following total/index scores will be evaluated as secondary endpoints: FACT-BL TOI (refer to as TOI), FACT-BL Total score, and NFBlSI-18 score.
  All the 5 subscales (PWB (0-28), FWB (0-28), EWB (0-24), SWB (0-28), and BlCS(0-48)) are summed as the FACT-BL total score (range 0-156), while the sum of PWB, FWB and BICS constitutes the FACT-BL TOI (range 0-104).
  NFBlSI-18 (range 0-72) is based on the scores of 16 items (GP4, C2, BL1, GP3, GE6, GE1, C6, BL5, GF5, GP2, GP1, GP6, C3, GP5, GF3, GF7) and 2 extra items "I feel weak all overall" and "I feel light-headed (dizzy)". The range of each item is 0-4.
  Higher score represent worse
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
Scores on a scale
  NFBLSI - 18 Score (Average overall visits): number analyzed (Participants) | 129 | 131 | 119
  NFBLSI - 18 Score (Average overall visits) | -3.9 (0.85) | -2.0 (0.87) | -5.7 (0.95)
  FACT-BL TOI (Average overall visits): number analyzed (Participants) | 129 | 131 | 119
  FACT-BL TOI (Average overall visits) | -5.8 (1.09) | -2.6 (1.11) | -8.0 (1.22)
  FACT-BL Total score (Average overall visits): number analyzed (Participants) | 129 | 131 | 119
  FACT-BL Total score (Average overall visits) | -8.0 (1.47) | -2.7 (1.51) | -10.1 (1.65)
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; NFBLSI- 18 score (Average overall visits); Test type: Superiority; p = 0.1373, Mixed Models Analysis — MMRM model included patient, treatment, cisplatin eligibility and visceral metastasis, visit and treatment by visit interaction as explanatory variables, and the appropriate baseline FACT-BL value as a covariate; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-0.6 to 4.36]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; NFBLSI- 18 score (Average overall visits); Test type: Superiority; p = 0.0034, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [1.26 to 6.27]
Statistical Analysis 3: Comparison: Combination Therapy vs Standard of Care; FACT-BL TOI (Average overall visits); Test type: Superiority; p = 0.1774, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-1.00 to 5.39]
Statistical Analysis 4: Comparison: Monotherapy vs Standard of Care; FACT-BL TOI (Average overall visits); Test type: Superiority; p = 0.0011, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [2.19 to 8.65]
Statistical Analysis 5: Comparison: Combination Therapy vs Standard of Care; FACT-BL Total score (Average overall visits); Test type: Superiority; p = 0.3494, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-2.27 to 6.38]
Statistical Analysis 6: Comparison: Monotherapy vs Standard of Care; FACT-BL Total score (Average overall visits); Test type: Superiority; p = 0.0011, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [2.96 to 11.71]

37. Secondary Outcome: Change From Baseline in FACT-BL (Derived NFBlSI-18 Score, FACT-BL TOI, and FACT-BL Total Score) by MMRM Analysis, PD-L1-Low/Negative Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: as for outcome 36
Time Frame: as for outcome 35
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
Scores on a scale
  NFBLSI - 18 Score (Average overall visits): number analyzed (Participants) | 91 | 73 | 69
  NFBLSI - 18 Score (Average overall visits) | -3.4 (1.01) | -3.8 (1.18) | -2.0 (1.16)
  FACT-BL TOI (Average overall visits): number analyzed (Participants) | 91 | 73 | 69
  FACT-BL TOI (Average overall visits) | -4.9 (1.18) | -5.0 (1.39) | -3.0 (1.36)
  FACT-BL Total score (Average overall visits): number analyzed (Participants) | 91 | 73 | 69
  FACT-BL Total score (Average overall visits) | -5.7 (1.62) | -6.5 (1.90) | -3.2 (1.86)
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; NFBLSI- 18 score (Average overall visits); Test type: Superiority; p = 0.3865, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-4.35 to 1.69]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; NFBLSI- 18 score (Average overall visits); Test type: Superiority; p = 0.2840, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-5.05 to 1.49]
Statistical Analysis 3: Comparison: Combination Therapy vs Standard of Care; FACT-BL TOI (Average overall visits); Test type: Superiority; p = 0.2970, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-5.41 to 1.66]
Statistical Analysis 4: Comparison: Monotherapy vs Standard of Care; FACT-BL TOI (Average overall visits); Test type: Superiority; p = 0.3026, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-5.85 to 1.83]
Statistical Analysis 5: Comparison: Combination Therapy vs Standard of Care; FACT-BL Total score (Average overall visits); Test type: Superiority; p = 0.3168, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-7.29 to 2.38]
Statistical Analysis 6: Comparison: Monotherapy vs Standard of Care; FACT-BL Total score (Average overall visits); Test type: Superiority; p = 0.2179, Mixed Models Analysis — [p-value comment as in outcome 36, analysis 1]; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-8.51 to 1.96]

38. Secondary Outcome: Improvement in Fatigue and Deterioration in Pain Per FACT-BL, Full Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: Fatigue will be based on the question of "I have a lack of energy" and pain will be based on the question of "I have pain", according to GP1 and GP4 in PWB, respectively.
  Improvement in fatigue is defined at least 1 point improvement from baseline using GP1 of FACT-BL.
  Deterioration in pain is defined as at least 1 point deterioration from baseline using GP4 of FACT-BL.
Time Frame: as for outcome 35
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 342 | 346 | 344
Participants
  Patients with improvement in fatigue: number analyzed (Participants) | 141 | 129 | 115
  Patients with improvement in fatigue | 38 | 37 | 24
  Patient with deterioration in pain: number analyzed (Participants) | 265 | 270 | 226
  Patient with deterioration in pain | 142 | 130 | 83
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Patients with improvement in fatigue; Test type: Superiority; p = 0.2419, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.8 to 2.6] — The OR and confidence interval (CI) were calculated using logistic regression, adjusting for PD-L1 status, visceral metastases and cisplatin eligibility status, with 95% CI calculated by profile likelihood
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Patients with improvement in fatigue; Test type: Superiority; p = 0.1553, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.9 to 2.8] — [estimate comment as in outcome 38, analysis 1]
Statistical Analysis 3: Comparison: Combination Therapy vs Standard of Care; Patient with deterioration in pain; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 2, 95% CI 2-sided [1.4 to 2.8] — [estimate comment as in outcome 38, analysis 1]
Statistical Analysis 4: Comparison: Monotherapy vs Standard of Care; Patient with deterioration in pain; Test type: Superiority; p = 0.0148, Regression, Logistic — [p-value comment as in outcome 18, analysis 1]; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.1 to 2.3] — [estimate comment as in outcome 38, analysis 1]

39. Secondary Outcome: Improvement in Fatigue and Deterioration in Pain Per FACT-BL, PD-L1-High Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: as for outcome 38
Time Frame: as for outcome 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 205 | 209 | 207
Participants
  Patients with improvement in fatigue: number analyzed (Participants) | 86 | 83 | 74
  Patients with improvement in fatigue | 23 | 24 | 14
  Patient with deterioration in pain: number analyzed (Participants) | 156 | 164 | 145
  Patient with deterioration in pain | 78 | 71 | 51
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Patients with improvement in fatigue; Test type: Superiority; p = 0.2473, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.7 to 3.4] — The OR and confidence interval (CI) were calculated using logistic regression, adjusting for visceral metastases and cisplatin eligibility status, with 95% CI calculated by profile likelihood
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Patients with improvement in fatigue; Test type: Superiority; p = 0.0148, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.8 to 3.8] — [estimate comment as in outcome 39, analysis 1]
Statistical Analysis 3: Comparison: Combination Therapy vs Standard of Care; Patient with deterioration in pain; Test type: Superiority; p = 0.0090, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.2 to 3.0] — [estimate comment as in outcome 39, analysis 1]
Statistical Analysis 4: Comparison: Monotherapy vs Standard of Care; Patient with deterioration in pain; Test type: Superiority; p = 0.1510, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.9 to 2.3] — [estimate comment as in outcome 39, analysis 1]

40. Secondary Outcome: Improvement in Fatigue and Deterioration in Pain Per FACT-BL, PD-L1-Low/Negative Analysis Set -Durvalumab + Tremelimumab Combination Therapy vs SoC and Durvalumab Mono Therapy vs SoC
Description: as for outcome 38
Time Frame: as for outcome 35
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
Number analyzed (Participants) | 137 | 137 | 137
Participants
  Patients with improvement in fatigue: number analyzed (Participants) | 55 | 46 | 41
  Patients with improvement in fatigue | 15 | 13 | 10
  Patient with deterioration in pain: number analyzed (Participants) | 109 | 106 | 81
  Patient with deterioration in pain | 64 | 59 | 32
Statistical Analysis 1: Comparison: Combination Therapy vs Standard of Care; Patients with improvement in fatigue; Test type: Superiority; p = 0.6763, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.5 to 3.2] — [estimate comment as in outcome 39, analysis 1]
Statistical Analysis 2: Comparison: Monotherapy vs Standard of Care; Patients with improvement in fatigue; Test type: Superiority; p = 0.6539, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.5 to 3.3] — [estimate comment as in outcome 39, analysis 1]
Statistical Analysis 3: Comparison: Combination Therapy vs Standard of Care; Patient with deterioration in pain; Test type: Superiority; p = 0.0092, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 2.2, 95% CI 2-sided [1.2 to 4.0] — [estimate comment as in outcome 39, analysis 1]
Statistical Analysis 4: Comparison: Monotherapy vs Standard of Care; Patient with deterioration in pain; Test type: Superiority; p = 0.0324, Regression, Logistic — [p-value comment as in outcome 19, analysis 1]; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.1 to 3.5] — [estimate comment as in outcome 39, analysis 1]

ADVERSE EVENTS:
Time Frame: From first administration of study treatment up to 90 days after last dose of study medication or date of initiation of the first subsequent therapy, whichever occurs first, approximately 5 years. All-cause mortality, from screening up to data cut-off date (27JAN2020, approximately 5 years).
Arm/Group | Combination Therapy | Monotherapy | Standard of Care
All-Cause Mortality (participants affected / at risk) | 255/342 | 263/346 | 270/344
Serious Adverse Events (participants affected / at risk) | 179/340 | 139/345 | 125/313
Other Adverse Events (participants affected / at risk) | 306/340 | 312/345 | 299/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=340) | Monotherapy (N=345) | Standard of Care (N=313)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (9) | 9 (9)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (4)
Haematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (4) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (3) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 5 (5) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 7 (7) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (8) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 16 (18) | 2 (2) | 4 (4)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (5) | 3 (3) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 4 (4)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 16 (19) | 6 (6) | 13 (13)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Listeriosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 15 (15) | 8 (9) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Prostatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 6 (7) | 6 (6)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 11 (11) | 4 (6)
Septic shock (Infections and infestations) | 3 (4) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 21 (26) | 17 (23) | 21 (28)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 7 (8) | 4 (4) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 6 (8)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 2 (2) | 2 (2)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 5 (5) | 8 (9)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 3 (3) | 2 (2) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 2 (2) | 2 (2)
Nephritis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary bladder rupture (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Penile haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 6 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=340) | Monotherapy (N=345) | Standard of Care (N=313)
Anaemia (Blood and lymphatic system disorders) | 51 (53) | 58 (63) | 163 (222)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 25 (50)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 89 (187)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 7 (10) | 47 (64)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 19 (22)
Hyperthyroidism (Endocrine disorders) | 21 (22) | 10 (10) | 1 (1)
Hypothyroidism (Endocrine disorders) | 31 (34) | 23 (23) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 41 (47) | 37 (50) | 27 (31)
Abdominal pain upper (Gastrointestinal disorders) | 19 (24) | 4 (4) | 8 (9)
Constipation (Gastrointestinal disorders) | 79 (88) | 66 (73) | 89 (113)
Diarrhoea (Gastrointestinal disorders) | 99 (146) | 63 (96) | 55 (78)
Dry mouth (Gastrointestinal disorders) | 23 (25) | 17 (18) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 12 (12) | 12 (14) | 18 (20)
Nausea (Gastrointestinal disorders) | 58 (65) | 74 (88) | 143 (237)
Vomiting (Gastrointestinal disorders) | 56 (66) | 36 (46) | 48 (61)
Asthenia (General disorders) | 54 (69) | 40 (49) | 68 (106)
Fatigue (General disorders) | 89 (106) | 98 (107) | 101 (127)
Malaise (General disorders) | 5 (5) | 4 (5) | 19 (21)
Oedema peripheral (General disorders) | 30 (39) | 36 (41) | 27 (33)
Pyrexia (General disorders) | 60 (80) | 50 (66) | 43 (63)
Nasopharyngitis (Infections and infestations) | 15 (16) | 18 (24) | 11 (13)
Urinary tract infection (Infections and infestations) | 54 (69) | 58 (82) | 46 (57)
Alanine aminotransferase increased (Investigations) | 14 (15) | 19 (21) | 21 (24)
Aspartate aminotransferase increased (Investigations) | 17 (18) | 15 (15) | 16 (21)
Blood alkaline phosphatase increased (Investigations) | 17 (18) | 20 (22) | 8 (10)
Blood creatinine increased (Investigations) | 17 (25) | 27 (33) | 31 (37)
Lipase increased (Investigations) | 23 (29) | 18 (33) | 4 (6)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 55 (135)
Platelet count decreased (Investigations) | 3 (3) | 4 (4) | 55 (124)
Weight decreased (Investigations) | 33 (34) | 21 (22) | 18 (18)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 29 (56)
Decreased appetite (Metabolism and nutrition disorders) | 72 (79) | 66 (74) | 80 (102)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (19) | 9 (12) | 10 (15)
Hyperkalaemia (Metabolism and nutrition disorders) | 17 (20) | 18 (24) | 18 (27)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (10) | 2 (2) | 21 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 (56) | 36 (45) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (38) | 41 (46) | 31 (34)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (21) | 25 (28) | 22 (23)
Dizziness (Nervous system disorders) | 27 (30) | 15 (21) | 25 (32)
Dysgeusia (Nervous system disorders) | 8 (9) | 10 (10) | 26 (30)
Headache (Nervous system disorders) | 20 (28) | 18 (18) | 16 (19)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 5 (5) | 16 (17)
Insomnia (Psychiatric disorders) | 25 (29) | 25 (25) | 14 (15)
Haematuria (Renal and urinary disorders) | 36 (40) | 39 (48) | 14 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (55) | 35 (41) | 18 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 30 (32) | 27 (30)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 23 (33)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 20 (23) | 5 (5) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (4) | 33 (33)
Pruritus (Skin and subcutaneous tissue disorders) | 93 (134) | 53 (71) | 14 (22)
Rash (Skin and subcutaneous tissue disorders) | 58 (77) | 30 (38) | 15 (18)
Hypertension (Vascular disorders) | 19 (20) | 19 (20) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT02516241/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT02516241/SAP_001.pdf